CLINICAL TRIAL: NCT01976468
Title: Metastases of Cutaneous Squamous Cell Carcinoma in Organ Transplant Recipients. The "SCOPE-ITSCC Metastases Study"
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Zurich (Other)
Collaborators: Leiden University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: SCOPE-ITSCC metastases
Record Dates: First submitted 2013-10-29; First posted 2013-11-05 (Estimated); Last update posted 2019-07-29 (Actual); Status verified 2019-07

CONDITIONS: Squamous Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Squamous Cell

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- SCC metastasis: organ transplant recipients
  Interventions: Other: SCC metastasis

INTERVENTIONS:
Other: SCC metastasis — occurrence of SCC metastasis

SUMMARY:
The investigators hypothesize that a low number of SCC in OTR will metastasize.

DETAILED DESCRIPTION:
In a large international multicenter prospective observational study a total number of 1000 OTR (organ transplant recipients) with a histologically proven cutaneous SCC (squamous cell carcinoma) will be included in 10 centers and followed during 2 years to establish the cumulative incidence of metastases in OTR with cutaneous SCC.

ELIGIBILITY:
Inclusion criteria:

* Organ-transplant recipients (OTR).
* Histologically proven cutaneous invasive SCC at time of inclusion

Exclusion criteria:

* Lack of consent.
* History of metastases of cutaneous SCC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: organ transplant recipients
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2013-11 (Actual); Primary Completion 2023-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
SCC metastasis detection | two years

CONTACTS AND LOCATIONS:
Overall Officials: Günther Hofbauer, Prof MD, Principal Investigator — University Hospital Zurich, Division of Dermatology; Jan Nico Bouwes Bavinck, Study Chair — Leiden University Medical Center; Roel Genders, MD, Study Director — Leiden University Medical Center
Locations (2):
- Leiden University Medical Center, Leiden, Netherlands
- University Hospital Zurich, Division of Dermatology, Zurich, Canton of Zurich, Switzerland